CLINICAL TRIAL: NCT07359872
Title: Relaxin Therapy for Atrial Fibrillation
Acronym: Relax-in-AF
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Deeptankar DeMazumder (U.S. Federal Agency)
Collaborators: Relaxera Pharmaceuticals (Unknown); McGowan Institute for Regenerative Medicine, University of Pittsburgh (Unknown); Relaxera Pharmazeutische Gesellschaft mbH & Co. KG (Unknown)
Responsible Party: Sponsor-Investigator, Deeptankar DeMazumder, Attending Physician in Cardiac Electrophysiology, VA Pittsburgh Healthcare System
Organization: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1923002
Record Dates: First submitted 2026-01-20; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation (AF); Arrhythmia; Oxidative Stress; Stroke; Major Cardiovascular Event; Heart Failure; Catheter Ablation; Ablation of Atrial Fibrillation
Keywords: randomized controlled crossover trial; Randomized clinical trial
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Stroke; Heart Failure | interventions — Relaxin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of care (including ablation) + Placebo x 9mo, then crossover to Relaxin therapy x 3mo (Experimental): Patients receiving the standard of care (which includes catheter ablation) will be treatment in a double blinded manner with (1) Placebo for the first 9 months; and then (2) Relaxin, instead of Placebo, for another 3 months.
  Interventions: Drug: Relaxin; Drug: Placebo
- Standard of care (including ablation) + Relaxin therapy x 9mo, then crossover to Placebo x 3mo (Experimental): Patients receiving the standard of care (which includes catheter ablation) will be treatment in a double blinded manner with (1) Relaxin for the first 9 months; and then (2) Placebo, instead of Relaxin, for another 3 months.
  Interventions: Drug: Relaxin; Drug: Placebo

INTERVENTIONS:
Drug: Relaxin — subcutaneous injections of Relaxin once daily
Drug: Placebo — subcutaneous injections of Placebo once daily

SUMMARY:
Atrial fibrillation (AF) is the most common heart rhythm disorder. The presence of AF increases the risk of death and is associated with a 5-6-fold increase in stroke incidence, due almost exclusively to thrombus formation in the heart. Current therapies for AF are limited. The evaluation of new, more effective treatments for preventing AF recurrence remains a critical unmet clinical need. AF is considered a progressive disease that increases in prevalence with age and can convert from "paroxysmal" to "persistent" to "permanent" AF in a single individual. This progression results, in part, from high oxidative stress and progressive adverse electrical changes in the heart. Compelling preclinical and clinical data indicate that Relaxin, a naturally occurring peptide hormone, may reverse the electrical remodeling. Thus, our overall objective is to investigate the effects of Relaxin in Veterans who have failed medical management for symptomatic AF and is referred to Cardiac Electrophysiology Laboratory for catheter ablation and pulmonary vein isolation. We will determine whether Relaxin therapy, in addition to the standard of care, counteracts the oxidative stress-related electrical derangement and reduces the post-ablation AF burden. A unique aspect of this proposal is that it is based in part on observations derived from the basic, translational and computational labs of the PI and co-investigators and from the observations by the PI while caring for patients with AF. As such, this proposal represents a true progression from the bench to the bedside. If successful, our findings may lead to the design of a new, more effective treatment for a major unmet public health problem in the United States as well as the world.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosed with AF and scheduled for elective catheter ablation for AF

Exclusion Criteria:

* Enrollment in another Greater than Minimal Risk Study
* Pregnant, nursing, or sexually active females not using birth control or having been surgically sterilized
* Females who plan to become pregnant during the trial period
* Patients diagnosed with "permanent" AF, complete heart block, or a reversible cause of AF (e.g., transient thyrotoxicosis)
* Patients that require antiarrhythmic medication to started or continued during and after the ablation procedure.
* Patients unable to tolerate Relaxin therapy or unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 390 days
  The Primary Safety Outcome includes the number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Ratio of the average daily AF burden before and after treatment | 390 days
  The Primary Efficacy Outcome includes the distribution of the ratio of the average daily AF burden before and after treatment over time. The daily AF burden is defined as the daily AF duration multiplied by the number of AF events including atrial ectopy.

CONTACTS AND LOCATIONS:
Overall Officials: Deeptankar DeMazumder, MD, PhD, Principal Investigator — (1) VA Pittsburgh Health System; (2) McGowan Institute for Regenerative Medicine.

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared as allowed by applicable VA, state, federal and IP rules and policies.
Supporting Information: Study Protocol
Time Frame: Data will be shared as allowed by applicable VA, state, federal and IP rules and policies.
Access Criteria: Data will be shared as allowed by applicable VA, state, federal and IP rules and policies.